CLINICAL TRIAL: NCT03203629
Title: Heart Sounds Registry In Patients Using The Wearable Cardioverter Defibrillator (HEARIT-Registry) Study Protocol
Brief Title: Heart Sounds Registry
Acronym: HEARIT-Reg
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0164
Record Dates: First submitted 2017-06-14; First posted 2017-06-29 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure; With Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Wearable Cardioverter Defibrillator (WCD) — Observe and compare the heart sound measurements recorded by the WCD
  Other Names: LifeVest; WCD

SUMMARY:
To conduct a prospective, observational study to evaluate the non-interventional feasibility of using heart sounds measurements recorded by the LifeVest® Wearable Cardioverter Defibrillator (WCD) for monitoring clinical evidence of heart failure decompensation.

DETAILED DESCRIPTION:
To conduct a prospective, observational study to evaluate the non-interventional feasibility of using heart sounds measurements recorded by the LifeVest® Wearable Cardioverter Defibrillator (WCD) for monitoring clinical evidence of heart failure decompensation.

Participants will be adult (age ≥ 18 years) heart failure patients with an ejection fraction (EF) ≤ 35% and eligible to wear the WCD for at least 3 months.

An FDA-approved WCD will be prescribed for at least 3 months of use after hospital discharge.

This is a multi-center, prospective, observational study.

The study will enroll a total of 300 subjects, anticipating that at least 250 subjects will complete the study. A maximum of 50 sites will enroll patients into the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed the WCD ≤ 10 days post-discharge after hospitalization with Heart Failure (HF), with and ischemic or non-ischemic cardiomyopathy.
* Patients who have an ejection fraction (EF) ≤ 35% at the time of WCD prescription.
* Patients are anticipated to wear the WCD for at least 3 months.
* The subject must be 18 years of age or older on the day of screening.

Exclusion Criteria:

* Patients with pacemakers, an implanted cardioverter defibrillator (ICD), or a cardiac resynchronization therapy device.
* Patients waiting for heart transplant.
* Patients with known evidence of atrial fibrillation on their most recent ECG recording.
* Patients currently hospitalized for acute myocardial infarction.
* Patients with a planned revascularization within 30 days of screening.
* Patients who are self-reporting to be pregnant.
* Patients participating in another clinical study.
* Patients not expected to live longer than 1 year.
* For patients in the United States, those who are unable or unwilling to provide written informed consent in English.
* For patients in Europe, those who are unable or unwilling to provide written informed consent in their country specific language or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adult (age ≥ 18 years) heart failure patients with an ejection fraction (EF) ≤ 35% and eligible to wear the WCD for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Observe the changes in the heart sounds measurement | 3 months
  Observe the changes in the heart sounds measurement (recorded by the WCD) with clinical evidence of heart failure decompensation during the three month WCD treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Szymkiewicz, MD, Study Director — Zoll Medical Corporation
Locations (33):
- United States (17):
  - MD Strategies Research Center, National City, California
  - JFK Medical Center, Atlantis, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Northside Hospital / Heart Institute, St. Petersburg, Florida
  - Carle Foundation Hospital, Urbana, Illinois
  - FRANCISCAN HEALTH Indianapolis, Indianapolis, Indiana
  - Cardiovascular Institute of Michigan, Clinton Township, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - Virtua The Cardiology Group, Moorestown, New Jersey
  - Virtua The Cardiology Group, Voorhees Township, New Jersey
  - Saratoga Clinical Research, Saratoga Springs, New York
  - MD First Research, Anderson, South Carolina
  - McLeod Regional, Florence, South Carolina
  - Chippenham Medical Center, Richmond, Virginia
  - West Virginia University Research, Morgantown, West Virginia
- Medizinische Universität Graz, Graz, Austria
- Germany (9):
  - Charité Berlin Benjamin Franklin, Berlin
  - Herzzentrum Dresden, Dresden
  - Uni Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Albertinenkrankenhaus HamburgKardiologie Albertinen-Krankenhaus, Hamburg
  - Asklepios St. Georg Hamburg, Hamburg
  - Sana Klinikum Hof,, Hof
  - Krankenhaus und MVZ Maria-Hilf Stadtlohn GmbH, Stadtlohn
  - University of Würzburg, Medizinische Klinik und Poliklinik I, Würzburg
- Poland (6):
  - American Heart of Poland S.A., Chrzanów
  - Wissmed Gdanskie Centrum, Gdansk
  - Klinika Elektrokardiologii Uniwersytetu Medycznego w Lodzi, Lodz
  - Spzoz Msw, Rzeszów
  - EMED Centrum Uslug Medycznych, Rzeszów
  - Wojewodzki Szpital Zespolony, Torun

IPD SHARING:
Plan to Share IPD: No